CLINICAL TRIAL: NCT07285655
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety and Efficacy of L606 (Treprostinil Liposome Inhalation Suspension) in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease (WHO Group 3)
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy L606 in Participants With PH-ILD
Acronym: Re-Spire
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L606-301
Record Dates: First submitted 2025-12-11; First posted 2025-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension Due to Lung Disease (Disorder)
Keywords: pulmonary hypertension; interstitial lung disease
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L606 (in combination with nebulizer) (Experimental)
  Interventions: Drug: L606
- Placebo (in combination with nebulizer) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L606 — L606 is a liposomal version of treprostinil intended for delivery via oral inhalation using a study issued nebulizer.
  Other Names: Treprostinil Liposome Inhalation Suspension
  Arms: L606 (in combination with nebulizer)
Drug: Placebo — Placebo will match L606 but contain no treprostinil.
  Arms: Placebo (in combination with nebulizer)

SUMMARY:
The purpose of this study is to find out if L606 is safe and if it helps people with high blood pressure in the lungs (pulmonary hypertension) caused by interstitial lung disease (PH-ILD, WHO Group 3). One of the main ways the study will check this is by seeing if people can walk further in six minutes (called the "six-minute walk test"). Another important (secondary) goal is to see how long it takes for PH-ILD to get worse while people are taking L606. One way the study will measure this is by looking at the distance people walk at different times in the study on different doses of L606. Throughout the study, doctors will also closely monitor for any side effects people have to make sure L606 is safe. People who decide to join this study will be randomly (like tossing a coin) placed into one of two groups: one group will get L606 and the other group will get a placebo, which will look like L606 but will not contain any active medicine. At the end of the initial blinded portion of the study, study participants may have the opportunity to enroll in an open-label extension portion of the study where all participants will receive L606.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between 18 years to 80 years old.
* Has a confirmed diagnosis of ILD based on High Resolution Computed Tomography (HRCT) chest imaging.
* Evidence of PH as demonstrated from Right Heart Catheterization (RHC) with the following hemodynamic parameters:
* Pulmonary vascular resistance (PVR) ≥ 320 dynes.sec/cm5 (i.e. 4 Woods Units (WU)), and
* Mean Pulmonary Artery Pressure (mPAP) of ≥ 25 mmHg, and
* - Pulmonary capillary wedge pressure (PCWP) or Left-Ventricular End Diastolic Pressure (LVEDP) of ≤ 15 mmHg.
* EV1/FVC (ratio) > 0.70.
* 6-minute walk distance ≥ 150 meters

Exclusion Criteria:

* PH in the updated WHO Classification Groups 1, 2, 4, or 5.
* Has evidence of clinically significant left-sided heart disease as defined by echocardiography.
* Participants with history of persistent/permanent or uncontrolled atrial fibrillation.
* Participants with severe obstructive sleep apnea.
* Has experienced exacerbation of underlying lung disease or active respiratory infection requiring antibiotics.
* Initiation of pulmonary rehabilitation.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6-minute walk distance (6MWD) as evaluated by the 6-minute walk test (6MWT) | 16 weeks

SECONDARY OUTCOMES:
Time to first occurrence of: -Death -Hospitalization due to a cardio-pulmonary indication related to underlying disease -Lung transplant -Decrease in 6MWD > 15% from Baseline related to disease under study at 2 consecutive visits >1 week apart | 24 weeks
Change from baseline in 6-minute walk distance (6MWD) as evaluated by the 6-minute walk test (6MWT) | 16 weeks
Change from baseline in 6-minute walk distance (6MWD) as evaluated by the 6-minute walk test (6MWT) | 24 weeks

IPD SHARING:
Plan to Share IPD: No